CLINICAL TRIAL: NCT03709979
Title: Inönü University Department of Anesthesia
Brief Title: Effect Of Position On Laryngeal Visualisation With The C-Mac Videolaryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zekine Begec, Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: C-Mac
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia; Intubation; Laryngoscopy
Keywords: video laryngoscopy; Pediatric patient; Position

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-MAC with folded towel position (Active Comparator): Children will be intubated by C-MAC videolaryngoscope with placing a folded towel under the shoulder.
  Interventions: Device: C-MAC videolaryngoscope
- C-MAC with flat position (Placebo Comparator): Children will be intubated by C-MAC videolaryngoscope with flat position (non-inserted a folded towel)
  Interventions: Device: C-MAC videolaryngoscope

INTERVENTIONS:
Device: C-MAC videolaryngoscope — An intubating device that is used for endotracheal intubation. Endotracheal intubation will be performed by anesthesiologist with C-MAC videolaryngoscope

SUMMARY:
The aim of this study is to demonstrate the effect of C-Mac videolaryngoscopy with Miller Blade size 0 and 1 on the intubation conditions in children less than 2 years age with a roll inserted under the shoulders.

DETAILED DESCRIPTION:
The laryngoscopic view of the glottis is improved when the angle of the line of vision between the pharyngeal - laryngeal axis and the oral cavity axis is narrow. A roll inserted under the shoulders of the infant will help line up the oral, laryngeal, and pharyngeal axes making direct laryngoscopy easier.

The investigators hypothesized that laryngoscopic view and intubation conditions using C-Mac videolaryngoscope with Miller Blade size 0 and 1 would be better with a roll under shoulder in children under 2 years.

ELIGIBILITY:
Inclusion Criteria:

* less than 2 years age undergoing general anaesthesia with tracheal intubation for elective surgery
* American Society of Anesthesiologists' physical status either 1 or 2 are included

Exclusion Criteria:

* upper respiratory tract infection within the previous 4 weeks
* airway difficulties in the preoperative evaluation
* unstable reactions during intubation

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Percentage of glottic opening score | immediately before endotracheal intubation
  Percentage of glottic opening score of 100% denotes visualization of the entire glottis, from the anterior commissure of the vocal cords to the inter-arytenoid notch. If no part of the glottic opening was visualized, the POGO score was recorded as 0%

SECONDARY OUTCOMES:
Time to intubation | From beginning of holding videolaryngoscope to seeing two meaningful end-tidal carbon dioxide levels up to 3 minutes
  Time to intubation will be measured from the time the videolaryngoscope entered the patient's mouth until the first capnograph trace is seen on the monitor

CONTACTS AND LOCATIONS:
Overall Officials: Zekine Begec, Professor, Principal Investigator — Inonu University Medical Faculty
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim EH, Lee JH, Song IK, Kim JT, Kim BR, Kim HS. Effect of head position on laryngeal visualisation with the McGrath MAC videolaryngoscope in paediatric patients: A randomised controlled trial. Eur J Anaesthesiol. 2016 Jul;33(7):528-34. doi: 10.1097/EJA.0000000000000448. PMID 26986776

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT03709979/Prot_SAP_000.pdf